CLINICAL TRIAL: NCT02079350
Title: Impact of %6 HES 130/0.4 and %4 Gelofusine Infusion on Kidney Function in the Living-donor Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Turkiye Yuksek Ihtisas Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, aslı demir, Associated professor, Turkiye Yuksek Ihtisas Education and Research Hospital
Other Study IDs: 11739
Record Dates: First submitted 2014-03-01; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Patients Undergoing Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- %4 Gelofusine: patients administered %4 Gelofusine during liver transplantation
  Interventions: Drug: %6 HES and %4 Gelofusine
- %6 HES: patients administered %6 HES during liver transplantation
  Interventions: Drug: %6 HES and %4 Gelofusine

INTERVENTIONS:
Drug: %6 HES and %4 Gelofusine

SUMMARY:
Although the negative impacts of colloid solutions with high molecular weight on renal functions, combination of lower molecular weight colloid varieties with crystalloid solutions and its use during intraoperative period have been subject to current research. Since the first liver transplantation, pre-or post-transplantation renal problems are still among the main causes of mortality and morbidity. The aim of the study was to evaluate the effects of fluid replacement solutions used intraoperatively on renal functions in elective living-donor liver transplantation.This study was approved by the Ethics Committee of Hospital and all patients were informed and gave written consent. Participants were patients scheduled for elective living-donor liver transplantation. Patients with normal renal function were randomly allocated to infusion with 6% HES 130/0.4 (HES Group) and 4% Gelofusine (GEL Group). Blood samples were obtained before induction of anesthesia (baseline), at the end of the operation, and postoperative days 1 and 4. Different eGFR formulas using creatinine (MDRD, CKD-EPI, and Cockraud Gault) were used to calculate estimated glomerular filtration rates.

ELIGIBILITY:
Inclusion Criteria:

-Normal kidney function

Exclusion Criteria:

* anormal kidney function
* cadaveric transplantation
* emergency operation
* patients less than 18 years old

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing living donor liver transplantation
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
renal dysfunction | 1 month

SECONDARY OUTCOMES:
mortality | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Turkey Yuksek Ihtisas Education and Research Hospital, Anesthesiology Clinic, Ankara, Turkey (Türkiye)